CLINICAL TRIAL: NCT00023972
Title: A Randomized, Open-Label, Multicenter Phase III Study Comparing the Efficacy and Safety of a Combination of Intravenous DX-8951f (Exatecan Mesylate) Plus Gemcitabine to Gemcitabine Alone in Patients With Locally Advanced or Metastatic Cancer of the Exocrine Pancreas Who Have Not Received Prior Chemotherapy
Brief Title: Gemcitabine With or Without Exatecan Mesylate in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068880; DAIICHI-8951A-PRT031; MSKCC-02011
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — exatecan; Gemcitabine

INTERVENTIONS:
Drug: exatecan mesylate
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if gemcitabine is more effective with or without exatecan mesylate in treating pancreatic cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of gemcitabine alone to that of gemcitabine and exatecan mesylate in treating patients who have locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with chemotherapy-naive locally advanced or metastatic cancer of the exocrine pancreas treated with exatecan mesylate and gemcitabine versus gemcitabine alone.
* Compare the measures of clinical benefit in patients treated with these regimens.
* Compare the anti-tumor efficacy of these regimens in this patient population.
* Determine the safety profile of exatecan mesylate and gemcitabine in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to performance status (60% vs 70-80% vs 90-100%), extent of disease (locally advanced vs metastatic), and prior radiotherapy for pancreatic cancer (yes or no). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive exatecan mesylate (DX-8951f) IV over 30 minutes immediately followed by gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive gemcitabine IV over 30 minutes once weekly for up to 7 weeks followed by one week of rest (course 1). For all subsequent courses, patients receive gemcitabine once weekly for 3 weeks followed by one week of rest. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly.

PROJECTED ACCRUAL: Approximately 340 patients (170 per treatment arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed epithelial cancer of the exocrine pancreas

  * Locally advanced (unresectable) or metastatic disease
* No islet cell tumor, lymphoma, or sarcoma of the pancreas
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 5 times ULN
* Albumin at least 2.8 g/dL

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No active congestive heart failure
* No uncontrolled angina
* No myocardial infarction

Other:

* No serious infection or life-threatening illness unrelated to tumor
* No other malignancy within the past 2 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No overt psychosis or incompetency that would preclude study
* No history of a positive serology for HIV
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior systemic anticancer immunotherapy for pancreatic cancer
* No concurrent anticancer immunotherapy or other biologic therapy

Chemotherapy:

* No prior systemic anticancer chemotherapy for pancreatic cancer
* Prior fluorouracil as a radiosensitizer allowed
* No prior gemcitabine as a radiosensitizer
* No other concurrent anticancer chemotherapy

Endocrine therapy:

* Concurrent megestrol for appetite stimulation allowed

Radiotherapy:

* At least 28 days since prior radiotherapy and recovered
* No prior radiotherapy to more than 25% of estimated bone marrow reserve
* No concurrent anticancer radiotherapy

Surgery:

* At least 28 days since prior major surgery and recovered
* No concurrent surgery for cancer

Other:

* No prior investigational or other systemic anticancer therapy for pancreatic cancer
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-07; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. DeJager, MD, FACP, Study Chair — Daiichi Sankyo
Locations (74):
- United States (66):
  - Intouch Research, Huntsville, Alabama
  - Providence Cancer Center, Mobile, Alabama
  - Arizona Clinical Research Center, Tucson, Arizona
  - Medical Oncology/Hematology, Gilroy, California
  - California Cancer Care, Inc., Greenbrae, California
  - Pacific Shores Medical Group, Long Beach, California
  - Cancer and Blood Institute of the Desert, Rancho Mirage, California
  - Sutter Cancer Center, Sacramento, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Medical Oncology and Hematology, P.C., Hamden, Connecticut
  - nTouch Research, Melbourne, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Peachtree Hematology and Oncology Consultants, P.C., Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - Central Georgia Hematology Oncology, P.C., Macon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Hope Center, Terre Haute, Indiana
  - Harbor Hospital Center, Baltimore, Maryland
  - Oncology-Hematology Associates, P.A., Clinton, Maryland
  - Providence Hospital Cancer Center, Southfield, Michigan
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - St. Joseph Oncology, Inc., Saint Joseph, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Midwest Hematology Oncology Consultants, Ltd., St Louis, Missouri
  - Billings Oncology Associates, Billings, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Nevada Cancer Center, Las Vegas, Nevada
  - Center for Cancer And Hematologic Disease, Cherry Hill, New Jersey
  - Hematology Oncology Associates, Morristown, New Jersey
  - Hematology and Oncology Group, Somerset, New Jersey
  - Summit Medical Group, P.A., Summit, New Jersey
  - HemOnCare, P.C., Brooklyn, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Nassau Hematology/Oncology PC, Lake Success, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - New York Medical College, Valhalla, New York
  - Buffalo Medical Group, P.C., Williamsville, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - N.W. Carolina Oncology & Hematology, P.A., Hickory, North Carolina
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Mid-Ohio Oncology/Hematology, Inc., Columbus, Ohio
  - Medical Oncology Associates of Wyoming Valley, P.C., Kingston, Pennsylvania
  - Lancaster Cancer Center, Lancaster, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Memorial Hospital Cancer Center - Chattanooga, Chattanooga, Tennessee
  - Williamson Medical Center, Franklin, Tennessee
  - Family Cancer Center, Germantown, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Sarah Cannon-Minnie Pearl Cancer Center, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Central Utah Medical Clinic, Provo, Utah
  - Intermountain Hematology/Oncology Associates, Inc., Salt Lake City, Utah
  - Rainier Oncology, Puyallup, Washington
  - Yakima Regional Cancer Care Center, Yakima, Washington
  - UW Cancer Center Wausau Hospital, Wausau, Wisconsin
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - Queen Elizabeth Hospital, PEI, Charlottetown, Prince Edward Island
  - CHUM Hopital Saint-Luc, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
- Veterans Affairs Medical Center - San Juan, San Juan, Puerto Rico

REFERENCES:
- [Result] Abou-Alfa GK, Letourneau R, Harker G, Modiano M, Hurwitz H, Tchekmedyian NS, Feit K, Ackerman J, De Jager RL, Eckhardt SG, O'Reilly EM. Randomized phase III study of exatecan and gemcitabine compared with gemcitabine alone in untreated advanced pancreatic cancer. J Clin Oncol. 2006 Sep 20;24(27):4441-7. doi: 10.1200/JCO.2006.07.0201. PMID 16983112